CLINICAL TRIAL: NCT04648410
Title: Administration of Systemic Corticosteroids Among Critically Ill Patients With COVID-19: Electronic Survey (ASAP-C Study)
Brief Title: Corticosteroids in Severe COVID-19(ASAP-C Study)
Acronym: ASAP-C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, assoc.prof.MD,Ph.D, Brno University Hospital
Other Study IDs: ASAP-C study
Record Dates: First submitted 2020-11-26; First posted 2020-12-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Severe COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Members of European Society of Intensive Care: Members of European Society of Intensive Care will obtain an electronic survey considering their routine clinical practice regarding the administration of systemic corticosteroids among patients with COVID-19 ARDS
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Members of European Society of Intensive Care will obtain an electronic survey considering their routine clinical practice regarding the administration of systemic corticosteroids among patients with COVID-19 ARDS
  Other Names: survey

SUMMARY:
Administration of systemic corticosteroids for patients with severe forms of severe acute respiratory syndrome(SARS-Co-2) infection are recommended by several guidelines. In the very beginning of SARS-Co-2 pandemic the early recommendation by professional organization was against routine use of corticosteroids for patients with coronavirus disease 2019 (COVID-19) acute respiratory distress syndrome (ARDS), despite previous data and clinical practice for patients with refractory or severe form of ARDS.

DETAILED DESCRIPTION:
Administration of systemic corticosteroids for patients with severe forms of SARS-Co-2 infection are recommended by several guidelines. In the very beginning of SARS-Co-2 pandemic the early recommendation by professional organization was against routine use of corticosteroids for patients with coronavirus disease 2019 (COVID-19) ARDS, despite previous data and clinical practice for patients with refractory or severe form of ARDS. But at the latest after publication of RECOVERY trial (Randomized Evaluation of Covid-19 Therapy, July 2020) and ensued metaanalysis of World Health Organization (WHO) working group, the routine administration of systemic corticosteroids was revisited. However, there are ongoing critical debate of the evidence regarding the dose, administration, timing and type of corticosteroids and ongoing randomized controlled trial (RCT) are challenging the recommendation of 6 mg of dexamethasone for all patients with severe form of COVID-19. The dynamic of COVID-19 surges, flip-flop of official recommendations within very short period of time and ongoing critical debate could be with possible variations of daily clinical practice regarding using systemic corticosteroids. In an electronic evaluation form that will be send to European Society of Intensive Care (ESICM) Members. The electronic survey will contain 10 question. In the questionnaire the participants will have to describe their routine clinical practice regarding administration of systemic corticosteroids among patients with COVID-19 ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Members of European Society of Intensive Care

Exclusion Criteria:

* not members of European Society of Intensive Care

Ages: 28 Days to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members of European Society of Intensive Care
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Systemic corticosteroids among patients with COVID-19 ARDS practice - questionnaire (electronic survey) | 1 month
  Administration of systemic corticosteroids among patients with COVID-19 ARDS practice in European countries - questionnaire (electronic survey)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Malaska, MD., Ph.D, Principal Investigator — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided